CLINICAL TRIAL: NCT00440726
Title: A Study of Bortezomib With Chemotherapy for Relapsed/Refractory Acute Lymphoblastic Leukemia
Brief Title: Bortezomib With Chemotherapy for Relapsed Pediatric Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T2005-003
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Pediatrics; Relapsed; Recurrence; Bortezomib; Velcade; Therapeutic Advances in Childhood Leukemia; Investigational; Childhood; ALL; Relapsed ALL; Refractory ALL; Relapsed pediatric ALL; Refractory pediatric ALL; TACL; Recurrent Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; pegaspargase; Doxorubicin; Cytarabine; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ph 1 Dose Escalation (Experimental): Intervention: Bortezomib with chemotherapy (dexamethasone, PEG-asparaginase, doxorubicin, cytarabine, methotrexate, and vincristine) and Triple IT therapy for patients who are CNS 2 or 3 at study entry. 3+3 escalation design.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Vincristine; Drug: Triple IT Therapy
- Ph 2 Efficacy and Safety (Experimental): Intervention: Bortezomib with chemotherapy (dexamethasone, PEG-asparaginase, doxorubicin, cytarabine, methotrexate, and vincristine) and Triple IT therapy for patients who are CNS 2 or 3 at study entry. Patients receive bortezomib at maximum tolerated dose (as established in the Phase 1 portion of the study) and are assessed for response and toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Vincristine; Drug: Triple IT Therapy

INTERVENTIONS:
Drug: Bortezomib — Intravenous on days 1, 4, 8 and 11. Dose assigned at study entry.
  Other Names: Velcade
Drug: Dexamethasone — 10 mg/m2/day divided BID, oral administration for 14 days.
  Other Names: Decadron
Drug: PEG-asparaginase — 2500 IU/m2/day, intramuscular injection on Days 2, 8, 15 and 22
  Other Names: Oncaspar
Drug: Doxorubicin — 60 mg/m2/day IV over 15 minutes on Day 1
  Other Names: Adriamycin; Rubex
Drug: Cytarabine — Given intrathecally on Day 1 of course 1 at the dose defined by age below.
  * 30 mg for patients age 1-1.99
  * 50 mg for patients age 2-2.99
  * 70 mg for patients >3 years of age
  Other Names: Cytosar-U; Ara-C; Arabinosylcytosine
Drug: Methotrexate — Given intrathecally to all patients who are CNS 1 at study entry on Day 15 at the dose defined by age below.
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  Other Names: Otrexup; Rasuvo; Rheumatrex; Trexall; Amethopterin
Drug: Vincristine — 1.5 mg/m2/dose IV push (maximum single dose 2 mg) on Days 1, 8, 15 and 22.
  Other Names: Oncovin; Leurocristine
Drug: Triple IT Therapy — Triple IT therapy will be given intrathecally on Day 8, 15, and 22 for patients who are CNS 2 and CNS 3 at study entry. Regimen/dosing as follows:
  Methotrexate-
  * <2 years: 8 mg
  * 2 - <3 y: 10 mg
  * 3 - <9 y: 12 mg
  * >=9 y: 15 mg
  Cytarabine:
  * <2 years: 16 mg
  * 2 - <3 y: 20 mg
  * 3 - <9 y: 24 mg
  * >=9 y: 30 mg
  Hydrocortisone:
  * <2 years: 8 mg
  * 2 - <3 y: 10 mg
  * 3 - <9 y: 12 mg
  * >=9 y: 15 mg

SUMMARY:
This is a Phase I/II study of a drug called bortezomib given in combination with chemotherapy drugs used to treat acute lymphoblastic leukemia (ALL) that has come back (recurred). Bortezomib is a drug that has been approved by the Food and Drug Administration (FDA) for treating adults with multiple myeloma which is a type of blood cancer. Bortezomib has been shown to cause cancer cells to die in studies done on animals (mice). Studies have been done that have shown that some adults and children with cancer have shown a response to bortezomib when it is used alone. Studies have also been done in adults to evaluate the dose of bortezomib that can be safely given in combination with other chemotherapy drugs.

DETAILED DESCRIPTION:
All patients will receive 1 course of chemotherapy unless medical complications prevent the administration of some of the drugs. Treatment will last about 1 month.

Treatment on this study will consist of a combination of 7 anti-cancer medications. The 7 anti-cancer medicines are bortezomib, vincristine, dexamethasone, PEG-asparaginase, doxorubicin, cytarabine (Ara-C), and methotrexate (MTX).

If you are in the Phase I portion of this study, you will be given an assigned dose of bortezomib. The dose of bortezomib will be based on doses given in previous studies done with adults and children. At each dose level of bortezomib, between 3 and 6 children will receive bortezomib in combination with chemotherapy. If the side effects are not too severe, the next group of children will receive a higher dose. The dose will continue to be increased until we find the dose that causes serious side effects. Your dose of bortezomib will not be increased. If you have bad side effects, your dose may be decreased.

The dose used during the Phase 2 part of this study will be determined by the outcome of the Phase I study. The highest dose used in Phase I that was tolerated without serious side effects will be the one used in Phase 2.

ELIGIBILITY:
Inclusion Criteria

The eligibility criteria listed below are interpreted literally and cannot be waived.

1. Age Patients must be < 21 years of age when originally diagnosed with ALL. Patient must be > 1 year of age at study entry.
2. Diagnosis Patients must have relapsed or refractory ALL with a M3 marrow (marrow blasts >25%). Patients with CNS I, II or III or testicular disease are eligible.
3. Performance Level Karnofsky > 50% for patients > 10 years of age and Lansky > 50% for patients < 10 years of age.
4. Prior Therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

   1. Prior anthracycline exposure: Patients must have less than 400mg/m2 lifetime exposure of anthracycline chemotherapy.
   2. Stem Cell Transplant (SCT): Patients are eligible after allogeneic stem cell transplant as long as patients are not actively being treated for graft-versus-host-disease (GvHD).
   3. Patients should not have received previous therapy using bortezomib (Velcdade® or PS-341).
   4. During the phase I portion of the trial, there is no limit on the number of prior treatment regimens. Patients with persistent disease after an induction attempt are eligible.
   5. During the phase II portion of the trial, patients must have had two or more prior therapeutic attempts defined as:

      * Persistent initial disease after two induction attempts, or
      * Relapse after one-reinduction attempt (2nd relapse), or
      * Persistent disease after first relapse and initial re-induction attempt

      (Patients in first relapse are not eligible for the phase II portion of the study)
   6. During the phase II portion of the trial, patients must have no more than 3 prior therapeutic attempts and it must be at least 3 months since the last treatment with a "VPLD" induction/re-induction regimen.
5. Reproductive Function

   1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
   2. Female patients with infants must agree not to breastfeed their infants while on this study.
   3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.

Exclusion Criteria

1. Drug Allergies

   Patients will be excluded if they have allergies to the following:
   * Asparaginase products
   * Boron
   * Mannitol
2. Renal Function Patients will be excluded if their serum creatinine is > 2 x the upper limit of normal for age at the institution's laboratory.
3. Liver/Pancreatic Function

   1. Direct bilirubin > 1.5x the institutional ULN for age. A total bilirubin result that is less than 1.5 times the institutional ULN for age may be used for eligibility if a direct bilirubin result is not available.
   2. SGPT (ALT) > 4 x institutional ULN
   3. Grade 3 or greater pancreatitis as defined by the CTCAE v3.0
   4. History of any L-asparaginase induced pancreatitis
   5. Amylase or Lipase > 2 x institutional ULN
4. Cardiac Function Patients will be excluded if their shortening fraction by echocardiogram is less than 30%.
5. Patients with Down Syndrome are excluded.
6. Infection

   * Patients will be excluded if they have an active uncontrolled infection.
   * Patients will be excluded if they have had a positive culture within 2 weeks of study entry.
7. Patients with grade 2 or greater motor or sensory neuropathy per CTC 3.0 criteria.
8. Patients planning on receiving other investigational agents while on this study. (An investigational agent is defined as any drug not currently approved for use in humans.)
9. Patients planning on receiving other anti-cancer therapies while on this study. Hydroxyurea for cyto-reduction is allowed prior to the start of therapy.
10. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
11. Patients who have started protocol therapy prior to enrollment. Patient may still enroll if IT therapy was given within 72 hours of study enrollment as part of the diagnostic lumbar procedure.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2006-08-04 (Actual); Primary Completion 2011-02-26 (Actual); Study Completion 2011-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Messinger, MD, Study Chair — Children's Hospital and Clinics of Minnesota
Locations (24):
- United States (20):
  - City of Hope, Duarte, California
  - Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Stanford University Medical Center, Palo Alto, California
  - UCSF School of Medicine, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami Cancer Center, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins / Sydney Kimmel Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - New York University Medical Center, New York, New York
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
- Universidade Federale de Sao Paulo/Hospital Sao Paulo, São Paulo, Brazil
- Sick Kids, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Messinger Y, Gaynon P, Raetz E, Hutchinson R, Dubois S, Glade-Bender J, Sposto R, van der Giessen J, Eckroth E, Bostrom BC. Phase I study of bortezomib combined with chemotherapy in children with relapsed childhood acute lymphoblastic leukemia (ALL): a report from the therapeutic advances in childhood leukemia (TACL) consortium. Pediatr Blood Cancer. 2010 Aug;55(2):254-9. doi: 10.1002/pbc.22456. PMID 20582937
- [Result] Messinger YH, Gaynon PS, Sposto R, van der Giessen J, Eckroth E, Malvar J, Bostrom BC; Therapeutic Advances in Childhood Leukemia & Lymphoma (TACL) Consortium. Bortezomib with chemotherapy is highly active in advanced B-precursor acute lymphoblastic leukemia: Therapeutic Advances in Childhood Leukemia & Lymphoma (TACL) Study. Blood. 2012 Jul 12;120(2):285-90. doi: 10.1182/blood-2012-04-418640. Epub 2012 May 31. PMID 22653976
- See also: Click here for more information about this protocol and the Therapeutic Advances in Childhood Leukemia Consortium — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 unique individual participants were enrolled into the study collectively for both Phase 1 and 2. The breakdown is as follows: 10 in the Phase I study and 21 in the Phase II study. There was, however, one patient that started on Phase I, Cohort 2 that was later eligible and rolled into the Phase II study.
Groups:
- Phase 1: Cohort 1 Bortezomib 1mg/m2/Day (Dose Level 1): The starting dose level of bortezomib will be 1 mg/m2/day given 2x week for 2 weeks on Days 1, 4, 8, and 11. The dose will be escalated to 1.3 mg/m2/day assuming that the maximum tolerated dose (MTD) is not exceeded. If the MTD is exceeded, the study will back down to the next whole dose level.
- Phase 1: Cohort 2 Bortezomib 1.3 mg/m2/Day (Dose Level 2): If the MTD is not exceeded at Dose Level 1, the next group of patients enrolled will escalate to Dose Level 2 of bortezomib at 1.3 mg/m2/day given on Days 1, 4, 8, and 11. This dose level is the highest possible dose level.
- Phase 2: Bortezomib 1.3 mg/m2/Day (Efficacy): After the MTD of bortezomib is defined with Phase 1, Phase 2 will enroll patients to receive bortezomib on Day 1, 4, 8 and 11 to evaluate activity of the regimen.
Period: Phase 1
Arm/Group | Phase 1: Cohort 1 Bortezomib 1mg/m2/Day (Dose Level 1) | Phase 1: Cohort 2 Bortezomib 1.3 mg/m2/Day (Dose Level 2) | Phase 2: Bortezomib 1.3 mg/m2/Day (Efficacy)
Started | 4 | 6 | 0
Completed | 3 | 5 | 0
Not Completed | 1 | 1 | 0
Not completed — Dose-Limiting Toxicity | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: Cohort 1 Bortezomib 1mg/m2/Day (Dose Level 1) | Phase 1: Cohort 2 Bortezomib 1.3 mg/m2/Day (Dose Level 2) | Phase 2: Bortezomib 1.3 mg/m2/Day (Efficacy)
Started | 0 | 0 | 22
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 31 unique individual participants were enrolled into the study collectively for both Phase 1 and 2. The breakdown is as follows: 10 in the Phase I study and 21 in the Phase II study. There was, however, one patient that started on Phase I, Cohort 2 that was later eligible and rolled into the Phase II study.
Groups:
- Phase 1 Dose Level 1: Bortezomib (Velcade): Intravenous on days 1, 4, 8 and 11, dose-escalation
  Dexamethasone: Intravenous or oral administration for 14 days.
  PEG-asparaginase: Intramuscular injection
  Doxorubicin: Intravenous infusion
  Cytarabine: Intrathecal administration on day 1
  Methotrexate: Intrathecal administration
  Vincristine: Intravenous push on days 1, 8, 15, 22
  The starting dose level of bortezomib will be 1 mg/m2/day given 2x week for 2 weeks on Days 1, 4, 8, and 11. The dose will be escalated to 1.3 mg/m2/day assuming that the maximum tolerated dose (MTD) is not exceeded. If the MTD is exceeded, the study will back down to the next whole dose level.
- Phase 1 Dose Level 2: If the MTD is not exceeded at Dose Level 1, the next group of patients enrolled will escalate to Dose Level 2 of bortezomib at 1.3 mg/m2/day given on Days 1, 4, 8, and 11. This dose level is the highest possible dose level
- Phase 2 Efficacy: After the MTD of bortezomib is defined with Phase 1, Phase 2 will enroll patients to receive bortezomib on Day 1, 4, 8 and 11 to evaluate activity of the regimen.
  Bortezomib (Velcade): Intravenous on days 1, 4, 8 and 11 at 1.3 mg/m2/day
  Dexamethasone: Intravenous or oral administration for 14 days.
  PEG-asparaginase: Intramuscular injection
  Doxorubicin: Intravenous infusion
  Cytarabine: Intrathecal administration on day 1
  Methotrexate: Intrathecal administration
  Vincristine: Intravenous push on days 1, 8, 15, 22
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 2 Efficacy | Total
Number analyzed (Participants) | 4 | 6 | 21 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 6 | 19 | 29
  Between 18 and 65 years | 0 | 0 | 2 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 7 | 15
  Male | 1 | 1 | 14 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 5 | 9
  Not Hispanic or Latino | 1 | 5 | 12 | 18
  Unknown or Not Reported | 0 | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 6 | 19 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Lineage [Count of Participants; unit: Participants] — Population: Patients in the dose escalation group were not stratified by lineage
  Participants
    number analyzed (Participants) | 0 | 0 | 21 | 21
    B-precursor ALL |  |  | 19 | 19
    T-cell ALL |  |  | 2 | 2
Prior Treatment Attempts [Count of Participants; unit: Participants]
  One | 1 | 4 | 0 | 5
  Two | 3 | 1 | 16 | 20
  Three | 0 | 0 | 5 | 5
  Four | 0 | 1 | 0 | 1
Previous Bone Marrow Transplant [Count of Participants; unit: Participants] — Population: Patients in the dose escalation group not stratified by previous BM transplant.
  Participants
    number analyzed (Participants) | 0 | 0 | 21 | 21
    None |  |  | 17 | 17
    Yes |  |  | 4 | 4
Bone Marrow M3 at study entry [Count of Participants; unit: Participants] — Population: Patients in the dose escalation group not stratified by leukemic blast status
  Participants
    number analyzed (Participants) | 0 | 0 | 21 | 21
    (all) |  |  | 21 | 21

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of a Dose-Limiting Toxicity (Phase 1)
Description: Toxicity will be graded using the CTCAE criteria, version 3.0. Dose-limiting toxicity will be defined as any of the following events that are deemed by the investigator as possibly, probably or definitely attributable to bortezomib: Grade 3 or 4 Sensory Neuropathy; Grade 3 or 4 Neuropathic pain (Neuralgia or peripheral nerve) lasting longer than 24 hours despite medical intervention; Marrow hypoplasia, which continues 6 weeks from the start of each course (less than 10% cellularity); and Grade 4 Non-Hematologic Toxicity excluding the following: Infection (septic shock, typhlitis), Fever/Neutropenia, Fatigue, Electrolyte abnormalities, Hyper/Hypoglycemia, Nausea or Vomiting, AST/ALT/Bilirubin elevations that return to grade 1 by the time of the next course.
Time Frame: Beginning with the first dose of investigational product until 30 days following the last dose of bortezomib
Measure: Count of Participants; unit: Participants
Groups:
- Ph 1, Dose Level 1 (1 mg/m2): Phase 1 patients receiving 1 mg/m2 dose of bortezomib
- Ph 1, Dose Level 2 (1.3 mg/m2): Phase 1 patients receiving 1.3 mg/m2 dose of bortezomib
Arm/Group | Ph 1, Dose Level 1 (1 mg/m2) | Ph 1, Dose Level 2 (1.3 mg/m2)
Number analyzed (Participants) | 4 | 6
Participants
  DLT | 0 | 1
  No DLT | 4 | 5

2. Primary Outcome: Achievement of Complete Remission (CR)
Description: * Complete Remission (CR): M1 (< 5% blasts) BM with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral counts (ANC>750/uL and platelet count >75 000/uL);
  * Complete Remission without Platelet Recovery (CRp): M1 BM with no circulating blasts or extramedullary disease and recovery of ANC (>750/uL) but insufficient recovery of platelets (<75 000/uL).
  * Partial Remission (PR): the disappearance of circulating blasts and achievement of M2 (5%-25% blasts) marrow status, without new sites of extramedullary disease, and with recovery of ANC (>750/uL).
  * Stable disease (SD): not satisfying the criterion for progressive disease (PD), or a recovery of ANC (>750/uL) but fails to qualify for CR, CRp, or PR.
  * Progressive Disease (PD): increase of at least 25% in the absolute number of circulating leukemia cells, development of new sites of extramedullary disease, or other lab or clinical evidence of PD, with or without recovery of ANC or platelets.
Time Frame: Day 29 of Course 1
Population: One Ph 1 patient received incorrect doses of Dexamethasone, so not evaluable for response. One Phase 2 patient achieved BM M1 but was treated with additional chemotherapy before peripheral recovery, so response to protocol treatment could not be evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Ph 1 Dose Escalation: Patients enrolled into the Phase 1 portion of the study
- Ph 2 B-Precursor ALL Patients: Patients enrolled into the Phase 2 portion of the study having B-Precursor ALL
- Ph 2 T-Cell ALL Patients: Patients enrolled into the Phase 2 portion of the study having T-Cell ALL
Arm/Group | Ph 1 Dose Escalation | Ph 2 B-Precursor ALL Patients | Ph 2 T-Cell ALL Patients
Number analyzed (Participants) | 9 | 19 | 2
Participants
  CR | 6 | 14 | 0
  CRp | 0 | 2 | 0
  SD/PD | 1 | 0 | 2
  BM-CR, CNS-SD | 1 | 0 | 0
  Death | 1 | 3 | 0

3. Post Hoc Outcome: Bone Marrow Response
Description: M1: Less than 5% blasts in a bone marrow aspirate and at least 200 cells counted.
  M2: 5-25% blasts in a bone marrow aspirate with at least 200 cells counted. M3: Greater than 25% blasts in a bone marrow aspirate with at least 200 cells counted.
Time Frame: Day 29 of Course 1
Population: All patients who enrolled and treated under Phase 2 will be evaluated at the end of Course 1 for treatment response as indicated by measure of bone marrow (M1, M2, or M3) or patient survival if death occurred.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 B-Precursor ALL Patients: Patients enrolled into the Phase 2 portion of the study having B-Precursor ALL
- Phase 2 T-cell ALL Patients: Patients enrolled into the Phase 2 portion of the study having T-Cell ALL
Arm/Group | Phase 2 B-Precursor ALL Patients | Phase 2 T-cell ALL Patients
Number analyzed (Participants) | 20 | 2
Participants
  M1 | 17 | 0
  M2/M3 | 0 | 2
  Death | 3 | 0

ADVERSE EVENTS:
Time Frame: 60 days, beginning with the first dose of investigational product until 30 days following the last dose of bortezomib
Description: The definition of adverse event used for data collection does not differ from that in the clinicaltrials.gov Definitions.
  For the purpose of reporting SAEs, all Grade 3 and 4 toxicities (CTCAE) are reported in this study record.
  Patients were evaluated regularly by the treating physician.
Groups:
- 1 mg/m2 Dose Group: Patients receiving a 1 mg/m2 dose of bortezomib (known as Dose Level 1 in the Phase 1 portion). All patients in this group were from the Phase 1 portion of the study.
- 1.3 mg/m2 Dose Group: Patients receiving a 1.3 mg/m2 dose of bortezomib (known as Dose Level 2 in the Phase 1 portion). This group includes patients from both the Phase 1 and Phase 2 portions of the study.
Arm/Group | 1 mg/m2 Dose Group | 1.3 mg/m2 Dose Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 5/27
Serious Adverse Events (participants affected / at risk) | 2/4 | 17/27
Other Adverse Events (participants affected / at risk) | 4/4 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/m2 Dose Group (N=4) | 1.3 mg/m2 Dose Group (N=27)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Bone marrow depression NOS (Blood and lymphatic system disorders) | 0 | 1
Caecitis (Gastrointestinal disorders) | 1 | 0
Cerebral ischaemia (Vascular disorders) | 0 | 2
Confusion (Psychiatric disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diarrhea NOS (Gastrointestinal disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Hyperglycemia NOS (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension NOS (Vascular disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Infection w/ Gr 3/4 ANC, Blood (Infections and infestations) | 1 | 8
Infection w/ Gr 3/4 ANC, Brain (Infections and infestations) | 0 | 1
Infection w/ Gr 3/4 ANC, Skin (Infections and infestations) | 0 | 1
Infection w/ norm ANC, Blood (Infections and infestations) | 0 | 1
Infection w/ unk ANC, Mucosa (Infections and infestations) | 0 | 1
Infection-Other (Infections and infestations) | 0 | 1
Lipase increased (Investigations) | 1 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophil count (Investigations) | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Platelet count decreased (Investigations) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/m2 Dose Group (N=4) | 1.3 mg/m2 Dose Group (N=27)
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 8
Activated partial thromboplastin time prolonged (Investigations) | 3 | 3
Alanine aminotransferase increased (Investigations) | 3 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 17
Blood alkaline phosphatase increased (Investigations) | 1 | 7
Blood amylase increased (Investigations) | 1 | 2
Blood bicarbonate decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 7
Blood creatinine increased (Investigations) | 0 | 4
Blood fibrinogen (Investigations) | 2 | 4
Clostridial infection NOS (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 6
Convulsions NOS (Nervous system disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cushingoid (Endocrine disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatology-Other (Skin and subcutaneous tissue disorders) | 0 | 2
Diarrhea NOS (Gastrointestinal disorders) | 3 | 8
Dizziness (Nervous system disorders) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Edema: limb (General disorders) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Fatigue (General disorders) | 0 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Hemoglobin (Blood and lymphatic system disorders) | 4 | 20
Headache (Nervous system disorders) | 1 | 2
Hepatobiliary/Pancreas-Other (Hepatobiliary disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 3 | 18
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 23
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 20
Hypoglycemia NOS (Metabolism and nutrition disorders) | 2 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 3 | 21
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 14
Hypotension NOS (Nervous system disorders) | 1 | 7
Hypothermia (General disorders) | 0 | 2
Implant site infection (Infections and infestations) | 1 | 0
Infection w/ Gr 3/4 ANC, Blood (Infections and infestations) | 0 | 2
Infection-Other (Infections and infestations) | 0 | 2
Leukopenia NOS (Blood and lymphatic system disorders) | 4 | 22
Lipase increased (Investigations) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5
Metabolic/Lab-Other (Investigations) | 0 | 2
Myalgia (General disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 8
Neutrophil count (Blood and lymphatic system disorders) | 4 | 12
Oral pain (Gastrointestinal disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain NOS (General disorders) | 0 | 3
Pain, External ear (General disorders) | 0 | 2
Pain-Other (General disorders) | 0 | 6
Pancreatitis NOS (Gastrointestinal disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3
Platelet count decreased (Blood and lymphatic system disorders) | 3 | 21
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 5
Rigors (General disorders) | 1 | 3
Sinus bradycardia (Cardiac disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 3
Tremor (Nervous system disorders) | 0 | 2
Vomiting NOS (Gastrointestinal disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days